CLINICAL TRIAL: NCT05570461
Title: Efficacy of Modified Constraint-Induced Movement Therapy on the Upper Limb Function of Sub-acute Stroke Patients in Peshawar Pakistan: A Randomized Controlled Trial
Brief Title: Efficacy of Modified Constraint-Induced Movement Therapy on the Upper Limb Function of Sub-acute Stroke Patients in Peshawar Pakistan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NCS University System (Other)
Responsible Party: Principal Investigator, Dr. Hazrat Bilal PT, Principal Invistigator, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU/IPMR/MS/22
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental group will receive Modified Constraint-Induced Movement Therapy and traditional physical therapy to the impaired upper limb based on the repetitive training of functional activities and behavioral shaping and a task-oriented approach, while the unaffected arm of subjects in the Modified Constraint-Induced Movement Therapy group will be constrained by wearing a mitten during the treatment session
  Interventions: Other: Modified Constraint-Induced Movement Therapy
- Control Group (Active Comparator): Control group therapy will consist of increasing upper limb function with the use of both hands. The session include active or active assistive range of motion exercises, unilateral and bimanual activities, balance and strength training or coordination exercises depending on the severity of motor impairment. Similar to group A, daily therapy will be conducted for 40 min/day, 6 days/ week for upto 2 weeks.
  Interventions: Other: Modified Constraint-Induced Movement Therapy

INTERVENTIONS:
Other: Modified Constraint-Induced Movement Therapy — Experimental group will receive Modified Constraint-Induced Movement Therapyand traditional physical therapy to the impaired upper limb based on the repetitive training of functional activities and behavioral shaping and a task-oriented approach, while the unaffected arm of subjects in the mCIMT group will be constrained by wearing a mitten during the treatment session and for 3 hours/day outside the therapy hours, 6(six) days/week for two weeks by an experienced Physical therapist.The time duration for Group A will be 40 minutes.

SUMMARY:
This RCT will also help the clinicians to provide the best treatment to their patients for better outcomes.

The objective of the study is to determine the efficacy of Modified Constraint-induced movement therapy on the Upper Limb function of Sub-acute stroke patients in Peshawar Pakistan.

Alternative Hypothesis: There will be a difference in the means of Modified Constraint-induced movement therapyand traditional physical therapy on the upper limb function of subacute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 30 to 60 years
* 2. Both female & male will be included.
* 3. Cognitive and lingual ability to communicate with the research staff.
* 4. A minimum of 10 degrees of active finger extension and 20 degrees of active wrist extension(16).
* 5. A history of a single stroke resulting in a hemiparesis

Exclusion Criteria:

* 1. Recurrent stroke during the training period.
* 2. Neurological or orthopedic disorders prohibiting the use of the paretic arm.
* 3. Patients who doesn't show willingness to participate in the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-11-04 (Estimated); Primary Completion 2023-08-12 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor function test | 4weeks
  Use mainly for post-stroke patients with impaired upper limb motor ability. The purpose of this test is to enumerate upper limb motor ability through a series of functional tasks. The WMFT is an instrument with high internal consistency, interrater reliability and test-retest reliability. The quality of movement during the task is measured by functional ability scale, a 6-point ordinal scale, where 0 = does not attempt with the impaired arm and 5 = arm movement appear to be normal.
  Higher the value higher will be the normal function.

IPD SHARING:
Plan to Share IPD: Undecided